CLINICAL TRIAL: NCT05969444
Title: The Impact of Endoscopic Surveillance of Atrophic Gastritis With and Without Intestinal Metaplasia on a High-risk Population for Gastric Cancer in Latin America: The ECHOS Cohort Study.
Brief Title: Endoscopic Surveillance on a High-risk Population for Gastric Cancer in Latin America: The ECHOS Cohort Study.
Acronym: ECHOS
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other); European Union (Other)
Responsible Party: Sponsor
Other Study IDs: 1230504 (AR)
Record Dates: First submitted 2023-06-28; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer; Dysplasia Stomach; Atrophic Gastritis; Helicobacter Pylori Infection
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Gastric mucosa biopsies were obtained following the USSBP as follows:
  * Two tissue samples obtained from the antrum (within 2 to 3 cm from the pylorus, from lesser and greater curvature)
  * One sample from the incisura angularis
  * Two samples from the body (one from lesser curvature, ~4 cm proximal from the angle,e and one from greater curvature, ~8 cm distal to cardia)
  * Samples from each anatomical location were collected either directed to a suspicious endoscopic finding of CAG or IM or following anatomical reference of the protocol if apparently normal gastric mucosa was visualized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the risk factors associated with incident HGD/GA in patients with CAG with or without IM who are enrolled in endoscopic surveillance, as well as to compare GA incidence according to the OLGA and OLGIM scales in patients 18 years or older.

. The main questions it aims to answer are:

* What risk factors are associated with incident HGD/GA in patients with CAG with or without IM?
* What is the comparative HGD/GA incidence according to the OLGA and OLGIM scales?

DETAILED DESCRIPTION:
The Endoscopic Cohort and Histological OLGA staging (ECHOS) study is a retrospective longitudinal cohort developed in the Pontificia Universidad Católica de Chile health care system, an open health care system with 3 endoscopic units in Santiago, Chile. Patients 18 years or older were eligible for the study if they had at least one non-urgent outpatient EGD with gastric biopsies collected following the USSBP between June 2015 and June 2021. The baseline EGD was defined as the earliest examination conducted between this time frame that met inclusion criteria. Participants were included in the cohort if they underwent a subsequent "surveillance" EGD. In order for the subsequent EGD to qualify as surveillance, it needed to occur at least 6 months after the baseline EGD and include gastric biopsies collected according to the USSBP; one exception to the USSBP requirement was if HGD or GA was detected on the surveillance (i.e. non-baseline) EGD. Patients with prior history of HGD or any type of gastric malignancy, gastrectomy or non-gastric active malignancy were excluded. Also, patients with HGD or GA on the baseline EGD were excluded. Patients with indefinite (IND) or low-grade dysplasia (LGD) on the baseline EGD were considered for the cohort.

ELIGIBILITY:
Inclusion Criteria:

* At least one non-urgent outpatient esophagogastroduodenoscopy (EGD) with gastric biopsies collected following the Updated Sydney System Biopsy Protocol (USSBP) between June 2015 and June 2021.
* Underwent a subsequent "surveillance" EGD. For the subsequent EGD to qualify as surveillance, it needed to occur at least six months after the baseline EGD and include gastric biopsies collected according to the USSBP; one exception to the USSBP requirement was if HGD or GA was detected on the surveillance.

Exclusion Criteria:

* Prior history of HGD or any type of gastric malignancy, gastrectomy, or non-gastric active malignancy.
* HGD or GA on the baseline EGD was excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients atteding an EGD at Pontificia Universidad Católica de Chile health care system, an open health care system with three endoscopic units in Santiago, Chile.
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
High grade dysplasia/Gastric adenocarcinoma | At least 6 months between first and second EGD, assessed up to 96 months
  Progression from chronic atrophic gastritis or intestinal metaplasia according to baseline Operative Link on Gastritis Assessment (OLGA) staging in baseline measurement to high-grade dysplasia and adenocarcinoma.
  The OLGA uses grades from in tiered scale from 0 to IV, resulting from the combination of atrophic changes (0 = absent; 1 = mild; 2 = moderate; 3 = severe) in the two mucosal compartments (antrum and corpus).

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Centro de especialidades médicas Marcoleta UC CHRISTUS, Santiago, Santiago Metropolitan
  - Centro Médico UC-CHRISTUS San Joaquín, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT05969444/Prot_SAP_000.pdf